CLINICAL TRIAL: NCT01601912
Title: Unraveling the Nature of Impaired Pain Inhibition in Patients With Chronic Whiplash-associated Disorders: a Randomized Controlled Clinical Trial for the Treatment of Central Sensitization
Brief Title: Unraveling the Nature of Impaired Pain Inhibition in Patients With Chronic Whiplash-associated Disorders
Status: Completed | Type: Observational
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Kelly Ickmans, MSc, Vrije Universiteit Brussel
Other Study IDs: WFWG-22
Record Dates: First submitted 2012-05-14; First posted 2012-05-18 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Whiplash Injuries
Keywords: Whiplash Injuries; Chronic Pain; Exercise; Cognition
MeSH Terms: conditions — Whiplash Injuries; Chronic Pain; Motor Activity | interventions — Atomoxetine Hydrochloride; Citalopram

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Atomoxetine NRI: We will modulate endogenous adrenergic pain inhibitory mechanisms by using a selective norepinephrine reuptake inhibitor (NRI).
  Interventions: Drug: Atomoxetine
- Citalopram SSRI: We will modulate serotonergic pain inhibitory mechanisms by using a selective serotonin reuptake inhibitor (SSRI)
  Interventions: Drug: Citalopram

INTERVENTIONS:
Drug: Atomoxetine — 40 mg, 1 application
  Other Names: Strattera (Eli Lilly Nederland B.V)
  Groups: Atomoxetine NRI
Drug: Citalopram — 20 mg, 1 application
  Other Names: Citalopram Sandoz (Sandoz N.V.)
  Groups: Citalopram SSRI

SUMMARY:
The primary study aim is to unravel the nature of impaired pain inhibition during exercise in patients with chronic Whiplash-Associated Disorders (WAD). This will be ascertained by examining whether activation of serotonergic and/or noradrenergic descending pathways improves pain inhibition during exercise in these patients. In addition, it is aimed at examining whether activation of serotonergic and/or noradrenergic descending pathways prevents post-exertional malaise following submaximal exercise in chronic WAD patients. A secondary study aim comprises of examining the effect of an acute submaximal exercise with and without activation of serotonergic or noradrenergic descending pathways on chronic WAD patients' cognitive performance. Furthermore, the isolated effect of activated serotonergic and noradrenergic descending pathways on chronic WAD patients' cognitive performance will be studied.

DETAILED DESCRIPTION:
Chronic Whiplash-Associated Disorders (WAD) is a debilitating, costly condition, and remains a challenge for clinicians, including physicians, rehabilitation specialists and physiotherapists. There is now consistent evidence for central sensitization in people with chronic WAD. In a previous study in chronic WAD patients, our group showed that pain inhibition during exercise is impaired and that a submaximal exercise triggers a severe relapse named post-exertional malaise. On the other hand, imbalance of serotonin (5-HT) and norepinephrine (NE) is likely to be responsible for malfunctioning of pain inhibitory pathways. Indeed, NE is required for activation of descending noradrenergic pathways with established nociceptive inhibitory properties. Serotonin reuptake inhibitor drugs activate serotonergic descending pathways that recruit, in part, opioid peptide-containing interneurons in the dorsal horn. It becomes more and more clear that the lack of pain inhibition accounts in part for various symptoms at rest and following exercise in particular (post-exertional malaise). However, the mechanisms behind the lack of pain inhibition during exercise remain to be revealed. Besides the lack of endogenous pain inhibition during exercise in people with chronic WAD, there appears to be sufficient evidence to support the presence of impaired cognitive function in chronic pain patients in general and preliminary evidence in chronic WAD patients in particular.

The present study aimed at examining whether activation of serotonergic and/or noradrenergic descending pathways improves pain inhibition during exercise in chronic WAD patients. In addition, it is aimed at examining whether activation of serotonergic and/or noradrenergic descending pathways prevents post-exertional malaise following submaximal exercise in these patients. A secondary study aim comprises of examining the effect of an acute submaximal exercise with and without activation of serotonergic or noradrenergic descending pathways on chronic WAD patients' cognitive performance. Furthermore, the isolated effect of activated serotonergic and noradrenergic descending pathways on chronic WAD patients' cognitive performance will be studied.We will modulate endogenous serotonergic and adrenergic pain inhibitory mechanisms by using a selective NE reuptake inhibitor (NRI) and a selective 5-HT reuptake inhibitor (SSRI). Endogenous pain inhibition and cognitive function (sustained and selective attention, and executive function) will be studied at rest and in response to exercise (1) under baseline condition, (2) after the intake of a NRI (Atomoxetine), and (3) after the intake of a SSRI (Citalopram).

ELIGIBILITY:
Inclusion Criteria for patients:

* WAD grades I to III according to the Quebec Task Force criteria
* experienced a whiplash trauma at least three months ago
* with chronic pain as a result of a whiplash injury
* 18-65 years of age and with Dutch as their native language will be able to participate

Exclusion Criteria for patients:

* other comorbidities or health issues that could explain the pain complaints
* < 18years > 65 years
* pregnant or until 1 year postnatal (for women)
* use of anti-depressive, anti-epileptic and pain medication.

Inclusion Criteria for healthy volunteers:

* 18-65 years of age and with Dutch as their native language will be able to participate
* having a sedentary job and doing < 3 h moderate physical activity/week
* being painfree without any chronic disease

Exclusion Criteria for healthy volunteers:

* < 18years > 65 years
* pregnant or until 1 year postnatal (for women)
* use of anti-depressive, anti-epileptic and pain medication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: WAD patients: primary care clinic & community sample Healthy people: community sample
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2013-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Changes in pain inhibition | Baseline before and after the submaximal graded exercise= day 1 A & B, after first intervention before and after the submaximal graded exercise= day 8 A & B, after second intervention before and after the submaximal graded exercise = day 15 A & B
  To investigate pain inhibition, a combination of temporal en spatial summation will be used on the example of Cathcart et al. (2009). Temporal summation is applied by using an analogue Wagner pressure algometer and spatial summation is induced by causing ischemic pain with an inflatable cuff.
Changes in psychomotor vigilance and alertness | Baseline before and after the submaximal graded exercise= day 1 A & B, after first intervention before and after the submaximal graded exercise= day 8 A & B, after second intervention before and after the submaximal graded exercise = day 15 A & B
  To investigate cognitive function we used the Psychomotor Vigilance Task (PVT) which is a 10-minute test.
Changes in selective attention and executive function | Baseline before and after the submaximal graded exercise= day 1 A & B, after first intervention before and after the submaximal graded exercise= day 8 A & B, after second intervention before and after the submaximal graded exercise = day 15 A & B
  The Stroop task is used to assess selective attention and executive function

SECONDARY OUTCOMES:
Change in scores on the Neck Disability Index questionnaire | Baseline = day 1, after the first intervention = day 8, after the second intervention = day 15
  The NDI was developed as a modification of the Oswestry Back Pain Index and was the first instrument designed to assess self-rated disability in patients with neck pain. The NDI is a valid and reliable instrument, sensitive to measure changes within a population of patients with neck pain.
Change in scores on the Brief Pain Inventory questionnaire | Baseline = day 1, after the first intervention = day 8, after the second intervention = day 15
  The BPI - short form includes 8 questions about one's pain levels and location in the body, and 7 questions about the daily interferences due to pain and it is sensitive to brief therapeutic interventions.
Changes in the scores on the Whiplash Associated Disorders Symptom list | Day 1 pre and post submaximal graded exercise and 24h after exercise = day 1 A,B&C, day 8 pre and post submaximal graded exercise & 24h after exercise = day 8 A,B&C, day 15 pre and post submaximal graded exercise & 24h after exercise = day 15 A,B&C
  This is a self-reported measure for assessing symptom severity in patients with WAD. The questionnaire is composed of the most reported WAD symptoms in the literature and some autonomic symptoms. Every symptom is presented by a visual analog scale (VAS) (100 mm), a method that is known for its validity and reliability.

CONTACTS AND LOCATIONS:
Overall Officials: Jo Nijs, PhD, Study Director — Vrije Universiteit Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Brussels, Brussels Capital, Belgium

REFERENCES:
- [Background] Van Oosterwijck J, Nijs J, Meeus M, Van Loo M, Paul L. Lack of endogenous pain inhibition during exercise in people with chronic whiplash associated disorders: an experimental study. J Pain. 2012 Mar;13(3):242-54. doi: 10.1016/j.jpain.2011.11.006. Epub 2012 Jan 24. PMID 22277322
- [Derived] Ickmans K, Malfliet A, De Kooning M, Goudman L, Hubloue I, Schmitz T, Goubert D, Aguilar-Ferrandiz ME. Lack of Gender and Age Differences in Pain Measurements Following Exercise in People with Chronic Whiplash-Associated Disorders. Pain Physician. 2017 Sep;20(6):E829-E840. PMID 28934789